CLINICAL TRIAL: NCT00053430
Title: Pharmacologic T Cell Costimulation In HIV Disease
Brief Title: Using the Drug Thalidomide to Stimulate T Cells in HIV-Infected People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01AI047742-01A1 (NIH); 7R01AI047742-02 (NIH)
Record Dates: First submitted 2003-01-29; First posted 2003-01-30 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: Immune Modulation; Thalidomide; Immune reconstitution; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Thalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Experimental): Participants will receive low dose thalidomide for 28 days
  Interventions: Drug: Thalidomide
- 2 (Placebo Comparator): Participants will receive low dose thalidomide placebo for 28 days
  Interventions: Drug: Thalidomide placebo

INTERVENTIONS:
Drug: Thalidomide — Tablet taken orally daily
  Arms: 1
Drug: Thalidomide placebo — Placebo tablet taken orally daily
  Arms: 2

SUMMARY:
Despite treatment with anti-HIV drugs, people infected with HIV continue to have problems with their immune systems. This study will evaluate whether the drug thalidomide, which stimulates the immune system's T cells, can improve immune system function in people with HIV.

DETAILED DESCRIPTION:
In patients with chronic HIV infection, HIV replication and abnormalities in immune function persist following treatment with highly active antiretroviral therapy (HAART). Specifically, costimulatory T cell interactions are impaired. The immune modulatory drug thalidomide was recently found to costimulate T cells. Pharmacologic T cell costimulation may compensate for the T cell deficiencies in people with HIV disease and improve immune function. This study will test whether thalidomide treatment enhances HIV and cytomegalovirus (CMV)-specific immunity in patients with HIV and CMV, and will evaluate the effect of thalidomide on HIV replication.

In this study, 40 HIV and CMV infected patients on HAART and 40 HIV uninfected CMV seropositive controls will be randomly assigned to low dose thalidomide or placebo treatment for 28 days. T cell responses and HIV replication and genetic diversification will be assessed.

ELIGIBILITY:
Inclusion Criteria

* HIV-infected for at least 5 years prior to study entry
* CD4 count of 300/mm3 or above
* Pre-HAART nadir CD4 count of 300/mm3 or less
* CMV infection
* HAART for 12 months prior to study entry
* Same effective HAART regimen for 3 months prior to study entry
* HIV viral load less than 200 copies/ml
* Clinically stable

Exclusion Criteria

* Active opportunistic infection
* Females of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-04; Primary Completion 2005-08 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Doubling in HIV Pol-specific CD8 cells, measured by ELISPOT | Through Day 28
Increase in CMV pp65 CD8 cells, measured by ELISPOT in the thalidomide treatment group | Throughout study
Increase in HIV p24-specific IFN-gamma-secreting CD4 cells in the thalidomide treatment group, measured by fluorescence-activated cell sorting (FACS) | Throughout study
Increase in cytomegalovirus (CMV)-specific interferon (IFN)-gamma-secreting CD4 T cells in the thalidomide treatment group, measured by FACS | Throughout study

SECONDARY OUTCOMES:
Increase in the frequency of keyhole limpet hemocyanin (KLH)-specific lymphocyte proliferative responses in the thalidomide treatment group | Throughout study
Increase in adverse events in the thalidomide treatment group | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Haslett, MD, Principal Investigator — Department of Microbiology and Immunology, University of Miami School of Medicine
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Background] Haslett PA, Hanekom WA, Muller G, Kaplan G. Thalidomide and a thalidomide analogue drug costimulate virus-specific CD8+ T cells in vitro. J Infect Dis. 2003 Mar 15;187(6):946-55. doi: 10.1086/368126. Epub 2003 Mar 6. PMID 12660941
- [Background] Haslett PA, Klausner JD, Makonkawkeyoon S, Moreira A, Metatratip P, Boyle B, Kunachiwa W, Maneekarn N, Vongchan P, Corral LG, Elbeik T, Shen Z, Kaplan G. Thalidomide stimulates T cell responses and interleukin 12 production in HIV-infected patients. AIDS Res Hum Retroviruses. 1999 Sep 1;15(13):1169-79. doi: 10.1089/088922299310269. PMID 10480630
- [Background] Matthews SJ, McCoy C. Thalidomide: a review of approved and investigational uses. Clin Ther. 2003 Feb;25(2):342-95. doi: 10.1016/s0149-2918(03)80085-1. PMID 12749503